CLINICAL TRIAL: NCT04408963
Title: VRC 611: A Phase 1 Safety and Pharmacokinetic Study to Evaluate a Human Monoclonal Antibody (mAb) VRC-HIVMAB0102-00-AB (CAP256V2LS) Administered Via Subcutaneous and Intravenous Injection in Healthy Adults
Brief Title: A Phase 1 Trial to Evaluate CAP256V2LS in Healthy Adults
Acronym: VRC 611
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200096; 20-I-0096
Record Dates: First submitted 2020-05-29; First posted 2020-06-01 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: HIV
Keywords: HIV Prevention; Broadly-Neutralizing Human Monoclonal Antibodies; First in Human; Anti-Drug Antibody Response; Antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: CAP256V2LS (5 mg/kg IV) (Experimental): CAP256V2LS (5 mg/kg) administered by intravenous (IV) infusion (Day 0)
  Interventions: Biological: VRC-HIVMAB0102-00-AB
- Group 2: CAP256V2LS (5 mg/kg SC) (Experimental): CAP256V2LS (5 mg/kg) administered by subcutaneous (SC) injection (Day 0)
  Interventions: Biological: VRC-HIVMAB0102-00-AB

INTERVENTIONS:
Biological: VRC-HIVMAB0102-00-AB — The VRC-HIVMAB0102-00-AB (CAP256V2LS) broadly neutralizing monoclonal antibody (bNAb) targets the V1V2 region of the HIV-1 envelope, is human in origin, and contains two amino acid modifications within the C-terminus of the heavy chain constant region designed to improve antibody half-life in vivo.
  Other Names: CAP256V2LS

SUMMARY:
Background:

HIV is a serious disease with no cure or vaccine to prevent it. Using antibodies could be a way to prevent HIV infection. Antibodies are made by the human body to fight germs. Researchers want to test an antibody, CAP256V2LS.

Objective:

To test CAP256V2LS to see if it is safe and how the body responds to it.

Eligibility:

Healthy people, ages 18-60

Design:

Participants were screened with a medical history, physical exam, and blood tests. Some females had a pregnancy test.

Participants were assigned to one of two groups. Based on their group, they got 1 dose of CAP256V2LS in 1 of 2 ways:

* Some participants got CAP256V2LS as an infusion. A thin tube was placed in an arm vein and CAP256V2LS was given into the vein using a pump.
* Some participants got CAP256V2LS injected under the skin. A small needle was used to inject CAP256V2LS into the fatty tissue of the belly, arm, or thigh. They got 1 to 4 injections.

On the day they got CAP256V2LS, participants gave blood samples at different time points.

Participants were asked to check their temperature every day for 7 days after receiving CAP256V2LS. They used a tool to measure any redness, swelling, or bruising they may have at the site where they received the study drug.

Participants had visits at least 2-3 times during the first week after they got CAP256V2LS. Then they had about 9 more visits over the next 6 months. Visits included blood tests.

DETAILED DESCRIPTION:
Design:

This open-label study evaluated CAP256V2LS (VRC-HIVMAB0102-00-AB) in healthy adults. The primary hypothesis was that subcutaneous (SC) and intravenous (IV) administrations of CAP256V2LS will be safe and well-tolerated in healthy adults. A secondary hypothesis was that CAP256V2LS will be detectable in human sera with a definable half-life.

Study Product:

The CAP256V2LS broadly neutralizing monoclonal antibody (bNAb) targets the V1V2 region of the HIV-1 envelope, is human in origin, and contains two amino acid modifications within the C-terminus of the heavy chain constant region designed to improve antibody half-life in vivo. This bNAb was developed by the VRC/NIAID/NIH in collaboration with The Centre for the AIDS Programme of Research in South Africa (CAPRISA) and is manufactured under current Good Manufacturing Practice (cGMP) regulations at the VRC Pilot Plant operated under contract by the Vaccine Clinical Materials Program (VCMP), Leidos Biomedical Research, Inc., Frederick. MD. The CAP256V2LS drug product is supplied at a concentration of 100 mg/mL in a sterile, aqueous, buffered solution of 6.25 mL in single-use 10 mL glass vials. R-Gene10 was added as a stabilizing agent to IV doses of CAP256V2LS. R-Gene10 (Arginine Hydrochloride Injection, USP) for intravenous infusion contains L-Arginine Hydrochloride, USP in Water for Injection (equivalent to a 10% solution).

Participants:

Healthy participants, 18-60 years of age

Study Plan:

This open-label study included 2 dosing regimens with CAP256V2LS administered at 5 mg/kg IV and 5 mg/kg SC. A single dose of the study product was administered on Day 0 as shown below.

VRC 611 Study Design

* Group 1

  * Study Product: CAP256V2LS
  * Participants per Group: 5
  * Dose (mg/kg) and Route Administered on Day 0: 5 mg/kg IV
* Group 2

  * Study Product: CAP256V2LS
  * Participants per Group: 5
  * Dose (mg/kg) and Route Administered on Day 0: 5 mg/kg SC

Total Participants: 10

Duration:

Study participation was approximately 24 weeks from the Day 0 product administration.

ELIGIBILITY:
* INCLUSION CRITERIA:

A volunteer must have met all of the following criteria to be included:

1. Able and willing to complete the informed consent process
2. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
3. Available for clinical follow-up through the last study visit
4. 18 to 60 years of age
5. Based on medical history and physical examination, in good health and without clinically significant findings within 84 days prior to enrollment.
6. Weight less than or equal to 115 kg
7. Willing to have blood samples collected, stored indefinitely, and used for research purposes

   Laboratory Criteria within 84 days prior to enrollment:
8. White Blood Cell (WBC) 2,500-12,000/mm^3
9. WBC differential either within institutional normal range or accompanied by the Principal Investigator (PI) or designee approval
10. Platelets = 125,000-500,000/mm^3
11. Hemoglobin within institutional normal range or accompanied by the PI or designee approval
12. Creatinine less than or equal to 1.1 x upper limit of normal (ULN) based on the institutional normal range
13. Alanine aminotransferase (ALT) less than or equal to 1.25 x ULN based on the institutional normal range
14. Negative for HIV infection by an FDA approved method of detection

    Criteria Specific to Women of Childbearing Potential:
15. Negative beta-human chorionic gonadotropin (HCG) pregnancy test (urine or serum) on day of enrollment, and prior to product administration
16. Agrees to use an effective means of birth control from at least 21 days prior to enrollment through the duration of study participation

EXCLUSION CRITERIA:

A volunteer was excluded if one or more of the following conditions applied:

1. Woman who is breast-feeding or planning to become pregnant during study participation
2. Any history of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis prior to enrollment that has a reasonable risk of recurrence during the study
3. Hypertension that is not well controlled
4. Receipt of any investigational study product within 28 days prior to enrollment. Note: SARS-CoV-2 vaccines approved by emergency use authorization are not exclusionary.
5. Receipt of any live attenuated vaccines within 28 days prior to enrollment.
6. Receipt of any vaccine within 2 weeks prior to enrollment/product administration
7. Prior receipt of a licensed or investigational monoclonal antibody
8. Prior receipt of an HIV vaccine
9. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a participant's ability to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Wu, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ko SY, Pegu A, Rudicell RS, Yang ZY, Joyce MG, Chen X, Wang K, Bao S, Kraemer TD, Rath T, Zeng M, Schmidt SD, Todd JP, Penzak SR, Saunders KO, Nason MC, Haase AT, Rao SS, Blumberg RS, Mascola JR, Nabel GJ. Enhanced neonatal Fc receptor function improves protection against primate SHIV infection. Nature. 2014 Oct 30;514(7524):642-5. doi: 10.1038/nature13612. Epub 2014 Aug 13. PMID 25119033
- [Background] Doria-Rose NA, Schramm CA, Gorman J, Moore PL, Bhiman JN, DeKosky BJ, Ernandes MJ, Georgiev IS, Kim HJ, Pancera M, Staupe RP, Altae-Tran HR, Bailer RT, Crooks ET, Cupo A, Druz A, Garrett NJ, Hoi KH, Kong R, Louder MK, Longo NS, McKee K, Nonyane M, O'Dell S, Roark RS, Rudicell RS, Schmidt SD, Sheward DJ, Soto C, Wibmer CK, Yang Y, Zhang Z; NISC Comparative Sequencing Program; Mullikin JC, Binley JM, Sanders RW, Wilson IA, Moore JP, Ward AB, Georgiou G, Williamson C, Abdool Karim SS, Morris L, Kwong PD, Shapiro L, Mascola JR. Developmental pathway for potent V1V2-directed HIV-neutralizing antibodies. Nature. 2014 May 1;509(7498):55-62. doi: 10.1038/nature13036. Epub 2014 Mar 2. PMID 24590074
- [Background] Doria-Rose NA, Bhiman JN, Roark RS, Schramm CA, Gorman J, Chuang GY, Pancera M, Cale EM, Ernandes MJ, Louder MK, Asokan M, Bailer RT, Druz A, Fraschilla IR, Garrett NJ, Jarosinski M, Lynch RM, McKee K, O'Dell S, Pegu A, Schmidt SD, Staupe RP, Sutton MS, Wang K, Wibmer CK, Haynes BF, Abdool-Karim S, Shapiro L, Kwong PD, Moore PL, Morris L, Mascola JR. New Member of the V1V2-Directed CAP256-VRC26 Lineage That Shows Increased Breadth and Exceptional Potency. J Virol. 2015 Oct 14;90(1):76-91. doi: 10.1128/JVI.01791-15. Print 2016 Jan 1. PMID 26468542
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-I-0096.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited for the study at the NIH Clinical Center in Bethesda, Maryland, USA.
Period: Overall Study
Arm/Group | Group 1: CAP256V2LS (5 mg/kg IV) | Group 2: CAP256V2LS (5 mg/kg SC)
Started | 5 | 5
Received Study Product | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Population included all enrolled participants. Weight represents weight at time of enrollment. Age represents age at enrollment day.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: CAP256V2LS (5 mg/kg IV) | Group 2: CAP256V2LS (5 mg/kg SC) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — Age represents age at enrollment day.
  years | 30.8 (10.0) | 41.4 (16.4) | 36.1 (14.0)
Age, Customized [Count of Participants; unit: Participants] — Age represents age at enrollment day.
  Participants
    21-30 years | 3 | 2 | 5
    31-40 years | 1 | 0 | 1
    41-50 years | 1 | 1 | 2
    51-60 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 1 | 3
  White | 1 | 4 | 5
  Multiracial | 2 | 0 | 2
  Hispanic/Latino | 1 | 2 | 3
  Non-Hispanic/Latino | 4 | 3 | 7
Weight (kg) [Mean (Standard Deviation); unit: kg] — Weight represents weight at time of enrollment.
  kg | 76.8 (20.0) | 68.8 (11.4) | 72.8 (15.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of CAP256V2LS Product Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Time Frame: 7 days after CAP256V2LS product administration, at approximately Week 1
Population: Population included all enrolled participants who received CAP256V2LS and provided safety data (via diary card).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: CAP256V2LS (5 mg/kg IV) | Group 2: CAP256V2LS (5 mg/kg SC)
Number analyzed (Participants) | 5 | 5
Participants
  Pain/Tenderness: None | 5 | 4
  Pain/Tenderness: Mild | 0 | 1
  Pain/Tenderness: Moderate | 0 | 0
  Pain/Tenderness: Severe | 0 | 0
  Pruritis (Itching): None | 5 | 4
  Pruritis (Itching): Mild | 0 | 1
  Pruritis (Itching): Moderate | 0 | 0
  Pruritis (Itching): Severe | 0 | 0
  Swelling: None | 5 | 4
  Swelling: Mild | 0 | 0
  Swelling: Moderate | 0 | 1
  Swelling: Severe | 0 | 0
  Redness: None | 5 | 2
  Redness: Mild | 0 | 1
  Redness: Moderate | 0 | 2
  Redness: Severe | 0 | 0
  Bruising: None | 5 | 5
  Bruising: Mild | 0 | 0
  Bruising: Moderate | 0 | 0
  Bruising: Severe | 0 | 0
  Any Local Symptom: None | 5 | 1
  Any Local Symptom: Mild | 0 | 2
  Any Local Symptom: Moderate | 0 | 2
  Any Local Symptom: Severe | 0 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of CAP256V2LS Product Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Time Frame: 7 days after CAP256V2LS product administration, at approximately Week 1
Population: Population included all enrolled participants who received CAP256V2LS and provided safety data (via diary card).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: CAP256V2LS (5 mg/kg IV) | Group 2: CAP256V2LS (5 mg/kg SC)
Number analyzed (Participants) | 5 | 5
Participants
  Malaise: None | 0 | 1
  Malaise: Mild | 2 | 1
  Malaise: Moderate | 3 | 2
  Malaise: Severe | 0 | 1
  Muscle Aches: None | 0 | 1
  Muscle Aches: Mild | 2 | 1
  Muscle Aches: Moderate | 3 | 2
  Muscle Aches: Severe | 0 | 1
  Headache: None | 0 | 2
  Headache: Mild | 2 | 0
  Headache: Moderate | 3 | 3
  Headache: Severe | 0 | 0
  Chills: None | 0 | 1
  Chills: Mild | 2 | 2
  Chills: Moderate | 3 | 1
  Chills: Severe | 0 | 1
  Nausea: None | 3 | 4
  Nausea: Mild | 0 | 1
  Nausea: Moderate | 2 | 0
  Nausea: Severe | 0 | 0
  Joint Pain: None | 1 | 3
  Joint Pain: Mild | 4 | 0
  Joint Pain: Moderate | 0 | 2
  Joint Pain: Severe | 0 | 0
  Temperature (Fever): None | 1 | 2
  Temperature (Fever): Mild | 2 | 0
  Temperature (Fever): Moderate | 2 | 3
  Temperature (Fever): Severe | 0 | 0
  Any Systemic Symptom: None | 0 | 1
  Any Systemic Symptom: Mild | 1 | 0
  Any Systemic Symptom: Moderate | 4 | 3
  Any Systemic Symptom: Severe | 0 | 1

3. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs) Following CAP256V2LS Product Administration
Description: Unsolicited adverse event (AE) data collection included AEs of all severities from the date of product administration through the Day 28 post-product administration visit. At other time periods greater than 4 weeks after the study product administration, only serious AEs (SAEs reported as a separate outcome and in the AE module) and new chronic medical conditions that required ongoing medical management (reported as a separate outcome) were recorded through the last study visit. The relationship between an AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 4 weeks after CAP256V2LS Product Administration
Population: Population included all enrolled participants who received CAP256V2LS and had safety data collected (via clinical assessment and/or lab results).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: CAP256V2LS (5 mg/kg IV) | Group 2: CAP256V2LS (5 mg/kg SC)
Number analyzed (Participants) | 5 | 5
Participants
  Related to Study Product | 5 | 3
  Unrelated to Study Product | 0 | 0
  Total Number of Participants who had One or More Non-Serious Unsolicited AE | 5 | 3

4. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Following CAP256V2LS Product Administration
Description: SAEs were recorded from receipt of study product administration through the last expected study visit at Week 24. The relationship between a SAE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 after CAP256V2LS product administration through the study participation, up to Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: CAP256V2LS (5 mg/kg IV) | Group 2: CAP256V2LS (5 mg/kg SC)
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

5. Primary Outcome: Number of Participants With New Chronic Medical Conditions Following CAP256V2LS Product Administration
Description: New chronic medical conditions that required ongoing medical management were recorded from receipt of first study product administration through the last expected study visit at Week 24. The relationship between a new chronic medical condition and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 after CAP256V2LS product administration through the study participation, up to Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: CAP256V2LS (5 mg/kg IV) | Group 2: CAP256V2LS (5 mg/kg SC)
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

6. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety Following CAP256V2LS Product Administration
Description: Abnormal laboratory results recorded as unsolicited adverse events (AEs) are summarized. Safety lab parameters included hematology (hemoglobin, hematocrit, mean corpuscular volume (MCV) platelets, and white blood cell (WBC), red blood cell (RBC), neutrophil, lymphocyte, monocyte, eosinophil and basophil counts) and chemistry (alanine aminotransferase (ALT) and creatinine). Complete Blood Count (CBC) with differential and Chemistry (ALT and creatinine) results were collected at different timepoints throughout the study per the protocol's schedule of evaluations. Comprehensive metabolic panel (CMP) was collected at baseline, and 2 weeks after product administration and as needed at additional timepoints. Institutional laboratory normal ranges as well as the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 were used.
Time Frame: Day 0 through 4 weeks after CAP256V2LS Product Administration
Population: Population includes all enrolled participants who received CAP256V2LS and had safety data collected via lab results.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: CAP256V2LS (5 mg/kg IV) | Group 2: CAP256V2LS (5 mg/kg SC)
Number analyzed (Participants) | 5 | 5
Participants
  ALT | 1 | 0
  Lymphocyte Count | 5 | 3
  Number of Participants with one or more Abnormal Laboratory Results AE Related to Study Product | 5 | 3
  Number of Participants with one or more Abnormal Laboratory Results AE Unrelated to Study Product | 0 | 0
  Total Number of Participants who had Any Abnormal Laboratory Results Reported as AEs | 5 | 3

7. Secondary Outcome: Pharmacokinetic (PK) Parameters of CAP256V2LS: Maximum Observed Serum Concentration (Cmax)
Description: Cmax is the peak serum concentration that CAP256V2LS achieves after it has been administered; it is determined as a maximum value on the summary pharmacokinetic (PK) curve for each study group.
Time Frame: Baseline through 24 weeks after CAP256V2LS product administration
Population: Population included participants who received CAP256V2LS (N=10).
Measure: Mean (Standard Deviation); unit: μg/ml
Arm/Group | Group 1: CAP256V2LS (5 mg/kg IV) | Group 2: CAP256V2LS (5 mg/kg SC)
Number analyzed (Participants) | 5 | 5
μg/ml | 155.57 (40.24) | 58.69 (8.64)

8. Secondary Outcome: Pharmacokinetic (PK) Parameters of CAP256V2LS: Time to Reach Maximum Observed Serum Concentration (Tmax)
Description: Tmax is the time it takes to reach Cmax of CAP256V2LS after it has been administered; it is determined based on the summary PK curve for each dose group.
Time Frame: Baseline through 24 weeks after CAP256V2LS product administration
Population: Population included participants who received CAP256V2LS (N=10).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1: CAP256V2LS (5 mg/kg IV) | Group 2: CAP256V2LS (5 mg/kg SC)
Number analyzed (Participants) | 5 | 5
days | 0.23 (0.35) | 6.32 (1.91)

9. Secondary Outcome: Pharmacokinetic (PK) Parameters of CAP256V2LS: Beta Half-life (T1/2b)
Description: Beta half-life (T1/2b) is the time required for half of the CAP256V2LS product to be eliminated from the serum.
Time Frame: Baseline through 24 weeks after CAP256V2LS product administration
Population: Population included participants who received CAP256V2LS (N=10).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1: CAP256V2LS (5 mg/kg IV) | Group 2: CAP256V2LS (5 mg/kg SC)
Number analyzed (Participants) | 5 | 5
days | 25.38 (2.47) | 27.00 (0.81)

10. Secondary Outcome: Pharmacokinetic (PK) Parameters of CAP256V2LS: Clearance Rate
Description: Clearance is the rate of CAP256V2LS elimination divided by the plasma CAP256V2LS concentration; determined based on the summary pharmacokinetic (PK) curve for each study group. Clearance following a SC administration is calculated as Clearance (CL)/Bioavailability (F).
Time Frame: Baseline through 24 weeks after CAP256V2LS product administration
Population: Population included participants who received CAP256V2LS (N=10).
Measure: Mean (Standard Deviation); unit: ml/day
Arm/Group | Group 1: CAP256V2LS (5 mg/kg IV) | Group 2: CAP256V2LS (5 mg/kg SC)
Number analyzed (Participants) | 5 | 5
ml/day | 84.32 (14.17) | 135.92 (8.89)

11. Secondary Outcome: Pharmacokinetic (PK) Parameters of CAP256V2LS: Volume of Distribution
Description: Theoretical volume that would be necessary to contain the total amount of administered drug at the same concentration as observed in plasma. It represents the degree to which a drug is distributed in body tissue rather than the plasma and calculated based in the PK curve for each study group. Volume of distribution following a SC administration is calculated as Volume of distribution (V)/Bioavailability (F).
Time Frame: Baseline through 24 weeks after CAP256V2LS product administration
Population: Population included participants who received CAP256V2LS (N=10).
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Group 1: CAP256V2LS (5 mg/kg IV) | Group 2: CAP256V2LS (5 mg/kg SC)
Number analyzed (Participants) | 5 | 5
Liter | 3.06 (0.34) | 5.29 (0.26)

ADVERSE EVENTS:
Time Frame: Unsolicited adverse event (AE) data collection included AEs of all severities from the date of product administration through the Day 28 post-product administration visit. At other time periods greater than 4 weeks after the study product administration, only serious AEs (SAEs) and new chronic medical conditions that required ongoing medical management (reported as a separate outcome) were recorded through the last study visit up to Week 24.
Description: Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment represent the number and percentage of participants reporting the event. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Arm/Group | Group 1: CAP256V2LS (5 mg/kg IV) | Group 2: CAP256V2LS (5 mg/kg SC)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: CAP256V2LS (5 mg/kg IV) (N=5) | Group 2: CAP256V2LS (5 mg/kg SC) (N=5)
Lymphopenia (Blood and lymphatic system disorders) | 5 | 3
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Transaminases Increased (Investigations) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 0 | 1
Administration site pain (General disorders) | 0 | 1
Administration site pruritus (General disorders) | 0 | 1
Administration site swelling (General disorders) | 0 | 1
Administration site erythema (General disorders) | 0 | 3
Malaise (General disorders) | 5 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Headache (Nervous system disorders) | 5 | 3
Chills (General disorders) | 5 | 4
Nausea (Gastrointestinal disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Pyrexia (General disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT04408963/Prot_SAP_ICF_001.pdf